CLINICAL TRIAL: NCT02555813
Title: Multicenter Non-interventional Study to Investigate Safety, Tolerability and Efficacy of Nab-paclitaxel in Clinical Routine Treatment of First-line Pancreatic Cancer Patients
Brief Title: Treatment of Pancreatic Cancer With Abraxane
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ABI-007-PANC-006
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer; nab-Paclitaxel; Gemcitabine; Non-interventional
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abraxane + Gemcitabine: Abraxane 125mg by intravenous( IV) infusion + Gemcitabine 1000mg by intravenous on Days 1, 8, 15 of every 21 day cycle until progression
  Interventions: Drug: Abraxane; Drug: Gemcitabine

INTERVENTIONS:
Drug: Abraxane — Abraxane By IV infusion on Days 1, 8, 15 and 28 until progression or toxicity
  Other Names: Nab-paclitaxel; ABI-007
Drug: Gemcitabine — Gemcitabine 1000mg IV infusion on Days 1, 8, 15 and 28 until disease progression or toxicity
  Other Names: Gemzar

SUMMARY:
This observational program collects data on tolerability, safety and efficacy regarding the use of Abraxane in metastatic pancreatic cancer patients in the daily clinical routine. Additionally data on dosage that is actually used in these patients will be collected. Patients who have pancreatic cancer and additional diseases can be documented in this study, too. Collected data might generate learnings on the optimal use of Abraxane in the daily routine setting.

DETAILED DESCRIPTION:
This observational program is aimed at gaining tolerability, safety and efficacy data with the routine use of Abraxane in its labeled indication in metastatic pancreatic cancer. Additionally data on real life dosing in daily clinical routine will be analyzed.

A detailed record of the medical history including co-morbidities and pre-treatment regimens will allow analysis of the impact thereof on tolerability, dosage and efficacy.

Hands-on experience with nab-paclitaxel is very limited in Austria and an non-interventional study could enhance knowledge on optimal drug handling and Adverse Event management.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic pancreatic carcinoma
2. Age > 18 years
3. Signed Informed Consent
4. Normal hepatic, renal and Bone Marrow functions

Exclusion Criteria:

1. Pregnant and lactating females 2. Previous treatment for metastatic pancreatic disease 3. Known hypersensitivity to nab-paclitaxel 4. Neutrophils < 1,5 x 10^9/L

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 5 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology.

SECONDARY OUTCOMES:
Best Overall Response | Up to 5 years
  Tumor response will be summarized as the percentage of participants who achieve a confirmed complete (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Voraberger, MD, Study Chair — Celgene Austria
Locations (19):
- Austria (19):
  - BHB Eisenstadt, Eisenstadt
  - LKH Feldkirch, Feldkirch
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - KH Elisabethinen Klagenfurt, Klagenfurt
  - LKH Klagenfurt, Klagenfurt
  - KH Krems, Krems
  - LKH Leoben, Leoben
  - KH Barmherzige Schwestern Linz, Linz
  - LKH Salzburg, Salzburg
  - LKH St. Pölten, Sankt Pölten
  - LKH Steyr, Steyr
  - Medical University Vienna, Vienna
  - KH St. Josephs, Vienna
  - KH Hanusch, Vienna
  - LKH Vöcklabruck, Vöcklabruck
  - Klinikum Wels, Wels
  - LKH Wr. Neustadt, Wiener Neustadt
  - KH Zams, Zams

REFERENCES:
- [Background] McBride A, Bonafede M, Cai Q, Princic N, Tran O, Pelletier C, Parisi M, Patel M. Comparison of treatment patterns and economic outcomes among metastatic pancreatic cancer patients initiated on nab-paclitaxel plus gemcitabine versus FOLFIRINOX. Expert Rev Clin Pharmacol. 2017 Oct;10(10):1153-1160. doi: 10.1080/17512433.2017.1365598. Epub 2017 Aug 21. PMID 28795609
- [Background] Kim S, Signorovitch JE, Yang H, Patterson-Lomba O, Xiang CQ, Ung B, Parisi M, Marshall JL. Comparative Effectiveness of nab-Paclitaxel Plus Gemcitabine vs FOLFIRINOX in Metastatic Pancreatic Cancer: A Retrospective Nationwide Chart Review in the United States. Adv Ther. 2018 Oct;35(10):1564-1577. doi: 10.1007/s12325-018-0784-z. Epub 2018 Sep 12. PMID 30209750
- [Background] Cartwright TH, Parisi M, Espirito JL, Wilson TW, Pelletier C, Patel M, Babiker HM. Clinical Outcomes with First-Line Chemotherapy in a Large Retrospective Study of Patients with Metastatic Pancreatic Cancer Treated in a US Community Oncology Setting. Drugs Real World Outcomes. 2018 Sep;5(3):149-159. doi: 10.1007/s40801-018-0137-x. PMID 29946913
- [Background] Young R, Mainwaring P, Clingan P, Parnis FX, Asghari G, Beale P, Aly A, Botteman M, Romano A, Ferrara S, Margunato-Debay S, Harris M. nab-Paclitaxel plus gemcitabine in metastatic pancreatic adenocarcinoma: Australian subset analyses of the phase III MPACT trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e325-e331. doi: 10.1111/ajco.12999. Epub 2018 Jun 22. PMID 29932294
- [Background] Fernandez A, Salgado M, Garcia A, Buxo E, Vera R, Adeva J, Jimenez-Fonseca P, Quintero G, Llorca C, Canabate M, Lopez LJ, Munoz A, Ramirez P, Gonzalez P, Lopez C, Reboredo M, Gallardo E, Sanchez-Canovas M, Gallego J, Guillen C, Ruiz-Miravet N, Navarro-Perez V, De la Camara J, Ales-Diaz I, Pazo-Cid RA, Carmona-Bayonas A. Prognostic factors for survival with nab-paclitaxel plus gemcitabine in metastatic pancreatic cancer in real-life practice: the ANICE-PaC study. BMC Cancer. 2018 Nov 29;18(1):1185. doi: 10.1186/s12885-018-5101-3. PMID 30497432
- [Background] Hegewisch-Becker S, Aldaoud A, Wolf T, Krammer-Steiner B, Linde H, Scheiner-Sparna R, Hamm D, Janicke M, Marschner N; TPK-Group (Tumour Registry Pancreatic Cancer). Results from the prospective German TPK clinical cohort study: Treatment algorithms and survival of 1,174 patients with locally advanced, inoperable, or metastatic pancreatic ductal adenocarcinoma. Int J Cancer. 2019 Mar 1;144(5):981-990. doi: 10.1002/ijc.31751. Epub 2018 Oct 3. PMID 30006989
- [Background] Barnes JA, Ellis ML, Hwang S, Emarine J, Merwin P, Salinas GD, Musher BL. Identification of Educational Gaps Among Oncologists Who Manage Patients with Pancreatic Cancer. J Gastrointest Cancer. 2019 Mar;50(1):84-90. doi: 10.1007/s12029-017-0033-8. PMID 29177608
- [Background] Woo W, Carey ET, Choi M. Spotlight on liposomal irinotecan for metastatic pancreatic cancer: patient selection and perspectives. Onco Targets Ther. 2019 Feb 21;12:1455-1463. doi: 10.2147/OTT.S167590. eCollection 2019. PMID 30863113
- [Background] Sonbol MB, Ahn DH, Goldstein D, Okusaka T, Tabernero J, Macarulla T, Reni M, Li CP, O'Neil B, Van Cutsem E, Bekaii-Saab T. CanStem111P trial: a Phase III study of napabucasin plus nab-paclitaxel with gemcitabine. Future Oncol. 2019 Apr;15(12):1295-1302. doi: 10.2217/fon-2018-0903. Epub 2019 Feb 15. PMID 30768369
- [Derived] Prager GW, Oehler L, Gerger A, Mlineritsch B, Andel J, Petzer A, Wilthoner K, Sliwa T, Pichler P, Winder T, Heibl S, Gruenberger B, Laengle F, Hubmann E, Korger M, Pecherstorfer M, Djanani A, Neumann HJ, Philipp-Abbrederis K, Woll E, Trondl R, Arnold-Schrauf C, Eisterer W. Comparison of nab-paclitaxel plus gemcitabine in elderly versus younger patients with metastatic pancreatic cancer: Analysis of a multicentre, prospective, non-interventional study. Eur J Cancer. 2021 Jan;143:101-112. doi: 10.1016/j.ejca.2020.11.003. Epub 2020 Dec 6. PMID 33296830